CLINICAL TRIAL: NCT06930404
Title: Innovation and Growth Network for Insightful Trends and Evaluation - Data Collection Study
Brief Title: Data Collection Study to Review Novel Methods for Diagnosing Obstructive Sleep Apnea
Acronym: Ignite
Status: Not yet recruiting | Type: Observational
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Other Study IDs: MA08042025
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Obstructive Sleep Apnea (OSA)
Keywords: diagnosis; screening
MeSH Terms: conditions — Sleep Apnea, Obstructive; Disease | interventions — Videotape Recording

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- People being investigated for obstructive sleep apnea: People who are undergoing testing (home sleep testing or polysomnography) due to suspicion of sleep apnea will be invited to take part
  Interventions: Other: facial scans, videos and heart rate variability measurements

INTERVENTIONS:
Other: facial scans, videos and heart rate variability measurements — Ignite app to collect data (videos, photos and heart rate variability)

SUMMARY:
This study will collect data on a range of signals such as facial scans, videos (including speaking, blinking and swallowing) and heart rate variability to assess whether any of these measures are useful for diagnosing obstructive sleep apnea

ELIGIBILITY:
Inclusion Criteria:

Adults aged >= 18 Ability to read and comprehend English

Exclusion Criteria:

* Previous diagnosis of OSA
* Respiratory diseases (such COPD, lung cancer, fibrosis of the lungs, lung injury)
* Subjects who are or may be pregnant, breastfeeding or within 6 weeks postpartum (which may impact HRV temporarily)
* Subjects with a pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults who are being tested for obstructive sleep apnea
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Correlation of measurement and obstructive sleep apnea status | 1 day
  - Area under the ROC curve (AUC) for each modality and their combinations in predicting moderate/severe OSA (AHI ≥15).

IPD SHARING:
Plan to Share IPD: Undecided